CLINICAL TRIAL: NCT05884502
Title: A Multicenter Prospective Randomized-controlled Interventional Study to Evaluate the Effect of High Dose Rosuvastatin Versus High Dose Rosuvastatin and Ezetimibe in Acute Ischemic Stroke Patients
Brief Title: A Multicenter Study to Evaluate the Effect of High Dose Rosuvastatin Versus Rosuvastatin and Ezetimibe in Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Yu, Sungwook, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021AN0073
Record Dates: First submitted 2023-04-10; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Dyslipidemias; Stroke, Acute Ischemic
MeSH Terms: conditions — Dyslipidemias; Ischemic Stroke | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Intervention Model Description: multicenter prospective randomized-controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination therapy (Experimental): combination of high-dose rosuvastatin and ezetimibe
  Interventions: Drug: combination of high-dose rosuvastatin and ezetimibe
- Single therapy (Active Comparator): high-dose rosuvastatin single administration group
  Interventions: Drug: high-dose rosuvastatin single administration

INTERVENTIONS:
Drug: combination of high-dose rosuvastatin and ezetimibe — combination of rosuvastatin 20mg and ezetimibe 10mg
  Arms: Combination therapy
Drug: high-dose rosuvastatin single administration — rosuvastatin 20mg monotherapy
  Arms: Single therapy

SUMMARY:
High-intensity statins are recommended for secondary prevention of stroke in patients with atherosclerotic ischemic stroke. According to the guidelines of the American Heart Association and the American Stroke Society, high-intensity or high-dose statins are recommended for high-risk groups of atherosclerotic cardiovascular disease (ASCVD). Statin therapy is recommended even if it is less than 100 mg/dL. The 2016 ESC/EAS and 2017 AACE guidelines include ischemic stroke and transient cerebral ischemic attacks caused by atherosclerosis in ASCVD, classifying them as ultra-high-risk groups, and recommending LDL cholesterol of less than 70 mg/dL as a treatment goal. The recently published guidelines for dyslipidemia in Korea also recommend that the target level of LDL cholesterol in patients with atherosclerotic ischemic stroke and transient ischemic attack be reduced to less than 70 mg/dL or 50% or more from the baseline.

According to a previous study on the efficacy and safety of high-intensity rosuvastatin in patients with ischemic stroke, it is not clear whether the use of rosuvastatin 20 mg prevents recurrence of cerebral infarction in the acute stage, but it is safe and effective for hemorrhagic conversion of cerebral infarction. In addition, the results were shown when rosuvastatin and ezetimibe were combined in patients with high cardiovascular risk, LDL cholesterol and total cholesterol decreased more in the combined group than in the single agent group. In a study comparing the group whose LDL cholesterol target was reduced to 70 mg/dL or less after stroke and the group maintained at 90-110 mg/dL, the group whose LDL cholesterol was controlled to 70 mg/dL or less It was confirmed that the incidence of cardiovascular disease was reduced. Existing studies aimed at general high-risk groups, not specific disease groups, and as in this study, studies were not conducted on a single disease group called acute stroke. In addition, there are only limited studies on the effectiveness and safety of diseases that occur mainly in the elderly, such as acute stroke. Therefore, there are currently no studies on the clinical efficacy and safety of high-intensity rosuvastatin and ezetimibe combination therapy for patients with acute cerebral infarction.

DETAILED DESCRIPTION:
Multicenter, randomized controlled trial to compare the efficacy and safety of the test group (high-dose rosuvastatin and ezetimibe combined administration group) and control group (high-dose rosuvastatin single administration group) to achieve the target LDL-C level in patients who have recently experienced an ischemic stroke; It is an open-label, investigator-led clinical trial.

In this clinical trial, treatment is performed according to the general treatment procedure for patients who have recently had an ischemic stroke. Subjects who agree to participate in the clinical trial and satisfy the selection and exclusion criteria are the test group (combination of high-dose rosuvastatin and ezetimibe). Administration group) and control group (high-dose rosuvastatin single administration group) are randomly assigned in a 1:1 ratio.

Clinical investigational drugs according to randomization are administered to hospitalized patients, and when discharged, they are allowed to take the provided clinical investigational drugs for a total of 90 days. After the baseline, on the 7th day or at discharge (1st follow-up), and on the 30th day (2nd follow-up), compliance with medication and occurrence of adverse reactions are observed, and on the 90th day (3rd follow-up), lipid concentration test is performed. Check LDL-C levels and compare with baseline LDL-C levels.

ELIGIBILITY:
Inclusion Criteria:

1. Those with primary hypercholesterolemia among those whose lesions were confirmed by brain CT or MRI within 48 hours of the onset of ischemic stroke
2. Adults 19 years of age or older
3. Patients who agreed to participate in this study

Exclusion Criteria:

1. Patients scheduled for carotid endarterectomy or stenting, cerebral artery stenting, coronary angioplasty and stenting, or coronary artery bypass surgery within 3 months
2. Patients with malignant tumors that have not been cured
3. Patients who have participated in other drug clinical trials within the last 30 days
4. Patients expected to experience side effects when taking rosuvastatin and ezetimibe
5. Patients who did not consent to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute value of LDL-C (low-density lipoprotein cholesterol) reduction | 90 days after enrollment
  low-density lipoprotein cholesterol reduction at 90 days after enrollment

OTHER OUTCOMES:
Percentage of reaching target LDL-C (low-density lipoprotein cholesterol) levels | 90 days after enrollment
  LDL-C (low-density lipoprotein cholesterol) < 70 mg/dL or 50% or more decrease from baseline
Changes in total cholesterol, HDL-C (high-density lipoprotein cholesterol), and TG (Triglyceride) levels at 3 months compared to randomization | 90 days after enrollment
  Changes in total cholesterol, HDL-C (high-density lipoprotein cholesterol), and TG (Triglyceride) levels at 90 days
Clinical event occurence- major cardiovascular adverse event (MACE) | 90 days after enrollment
  MACE; relapse of stroke, cardiovascular death, other death, occurrence of coronary artery disease, occurrence of myocardial infarction requiring percutaneous coronary intervention
Clinical Stroke Scale | 90 days after enrollment
  NIHSS (National Institute of Health stroke scale) score,
Clinical Stroke Scale | 90 days after enrollment
  mRS (modified Rankins scale) score
Safety endpoints | 90 days after enrollment
  newly diagnosed diabetes mellitus
Safety endpoints | 90 days after enrollment
  newly developed muscle symptoms measured with statin related muscle symptoms questionnaire (SAMS-Q)
Safety endpoints | 90 days after enrollment
  liver enzyme levels (AST in IU/L, ALT in IU/L)
Safety endpoints | 90 days after enrollment
  development of intracranial hemorrhage

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Koera University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No